CLINICAL TRIAL: NCT05488080
Title: PAINED: Project Addressing INequities in the Emergency Department
Acronym: PAINED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Monika Goyal, Associate Professor of Pediatrics and Emergency Medicine, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FP00005944 / 1R61DK135406 - 01
Record Dates: First submitted 2022-07-15; First posted 2022-08-04 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Pain; Appendicitis; Bias, Racial; Fractures, Bone
MeSH Terms: conditions — Pain; Appendicitis; Racism; Fractures, Bone

STUDY DESIGN:
Intervention Model Description: The study design is a pragmatic clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Department-level audit and feedback and electronic health record-embedded clinical decision support (Experimental): Clinicians will receive monthly pooled, department-level 'Equity Report Cards' that will provide aggregate information on clinical data stratified by patient race/ethnicity. Subsequently, for all visits that may be related to appendicitis or long bone fracture, clinicians will then receive real-time, electronic health record-embedded clinical decision support regarding pain management.
  Interventions: Behavioral: Department-level audit and feedback and electronic health record-embedded clinical decision support

INTERVENTIONS:
Behavioral: Department-level audit and feedback and electronic health record-embedded clinical decision support — This intervention will provide clinicians with Equity Report Cards and clinician decision support on mitigating disparities in quality of care.

SUMMARY:
Racial and ethnic inequities in health care quality have been described across a broad range of clinical settings, patient populations, and outcomes. Our overarching goal is to eradicate health care inequities through evidence-based interventions. The objectives of this proposal are to develop and test the impact of two interventions on overcoming clinician implicit bias and mitigating inequities in the management of pain among children seeking care in the emergency department for the treatment of appendicitis or long bone fractures.

ELIGIBILITY:
Inclusion Criteria:

* All Children's National Hospital Emergency Department clinicians
* Patients 0-21 years with symptoms suggestive of appendicitis or long bone fracture

Exclusion Criteria:

* Emergency Severity Index (ESI 1)

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22032 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2026-08-23 (Estimated); Study Completion 2026-08-23 (Estimated)

PRIMARY OUTCOMES:
Pain reduction | Equity Report Cards provided monthly to clinicians over a 24-month period
  Percentage of patients with pain reduction, pain is measured on a 0 to 10 scale, 0 is the minimum and 10 is the maximum, a lower score is a better outcome.
Analgesia use | Equity Report Cards provided monthly to clinicians over a 24-month period
  Rate of analgesia use

CONTACTS AND LOCATIONS:
Overall Officials: Monika Goyal, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No